CLINICAL TRIAL: NCT07235631
Title: Exergames Enjoyment Using Various Devices and Awareness of Their Use for Physical Activity and Health Improvement Among Young Adults
Brief Title: Exergames Enjoyment and Awareness of Their Use for Physical Activity and Health Among Young Adults
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Magdalena Cyma-Wejchenig, Principal Investigator, Poznan University of Physical Education
Other Study IDs: 220/23
Record Dates: First submitted 2025-10-02; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy Young Adults
Keywords: Exergames; Physical activity promotion; Virtual reality; Exercise enjoyment; Gamification; Digital health technologies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy volunteers (university students, age 18-36): Single cohort of healthy volunteers (university students, age 18-36), all of whom were exposed to multiple exergame devices in a single laboratory session

SUMMARY:
The goal of this observational, non-interventional study is to explore how different exergame devices are perceived by young adults in terms of enjoyment and awareness of their potential use for physical activity and health improvement. Participants are exposed to several commercially available exergame systems in a standardized laboratory setting, with no intention to modify their health, fitness, or behavior.

The main questions it aims to answer are:

* Do different exergame devices provide different levels of enjoyment (as measured by the Exergame Enjoyment Questionnaire)?
* How do young adults perceive the usefulness of various exergames for supporting physical activity and health?

Participants will:

* Complete a brief questionnaire on physical activity habits.
* Take part in short (about 10 minutes each) exposure sessions using different exergame devices (VR, Wii Fit, Dance platform, Ring Fit) - approximately 50 minutes in total per participant.
* Be randomly assigned to complete post-exposure questionnaires referring to one randomly selected device only.

No interventions are applied and no pre-post measurements are collected; the study is purely observational, focusing on subjective user experience rather than behavioral or physiological change.

DETAILED DESCRIPTION:
This study investigates exergames as interactive digital technologies that combine gaming elements with physical activity. The research focuses on multiple commercially available devices representing different modes of interaction (virtual reality, motion sensors, balance platforms, and handheld controllers). The design followed a cross-sectional, single-session observational approach with a single sample of healthy young adults.

All participants completed baseline self-reports on physical activity, followed by standardized, non-interventional exposure to several exergame devices. Each participant interacted with all devices in an assigned order, under controlled laboratory conditions, with no manipulation intended to modify physical fitness, health status, or behaviour.

The exposure served solely for observational and comparative purposes to collect subjective evaluations rather than to test any training or therapeutic effects. Outcomes (structured evaluations regarding enjoyment and perceived utility of each exergame) were collected immediately post-exposure only, with no pre-post measurements or longitudinal follow-up.

Five commercially available exergame systems were included to represent diverse interaction modes:

* Sony PlayStation 4 with PlayStation VR (PS VR), using immersive virtual reality headsets with motion tracking.
* Nintendo Wii Fit, employing a balance board platform to capture weight shifts and postural control.
* Dance Revolution (DDR/StepMania-type system), based on a floor platform interface for rhythm-based movement.
* Nintendo Switch with Ring Fit Adventure (RFA), combining a resistance ring and leg strap for sensor-based motion detection.
* Meta Quest 2 (standalone VR headset), providing fully immersive virtual environments with handheld controllers.

All devices were used in a standardized observation setting (10-minute exposure per device, total 50 minutes per participant) with consistent instructions across participants. The sequence of device use was randomized to minimize order effects but not to assign participants to different intervention arms.

After completing all exposures, participants were randomly assigned to complete post-exposure questionnaires referring to one exergame device only. This procedure ensured that each participant evaluated a single system in detail, while overall responses were distributed evenly across all devices.

The study applied validated psychometric tools (Exergame Enjoyment Questionnaire, EEQ) as the primary outcome measure, alongside a custom survey assessing perceived training potential, engagement, and expected health benefits. All variables represent subjective, self-reported outcomes collected in a single measurement session.

Statistical analyses (non-parametric tests such as Kruskal-Wallis with post-hoc comparisons) examined differences in enjoyment ratings across devices. Descriptive analyses summarized participants' responses regarding device preferences, awareness of exergame applications, and prior experience.

This study does not test any health-related intervention, treatment, or behavioral modification. It is an observational, exposure-only investigation designed to explore user experience and perception of different exergame modalities, without inducing or evaluating physiological or functional change.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older,
* proficient in verbal communication,
* fully mobile.

Exclusion Criteria:

* any health conditions that could affect reaction time or PA levels, such as neurological disorders,
* current injuries,
* pain affecting the spine or upper limbs.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students of Poznan University of Physical Education
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Enjoyment during exergame play | EEG was assessed immeditely afterwards exergaming session
  Tool:
  Exergame Enjoyment Questionnaire (EEQ) - validated 20-item instrument which integrates elements from the Game Engagement Questionnaire (GEQ), the Intrinsic Enjoyment Questionnaire (IEQ), and items from the PA Enjoyment Scale (PACES).
  The questionnaire captures multiple aspects of enjoyment, including emotional engagement, immersion, perceived physical benefits, and control, as well as potential negative experiences such as frustration or physical discomfort.
  Number of items: 20;
  Scoring:
  Likert scale (in range 1-5), with higher values indicating greater enjoyment; subscales were aggregated to provide an overall enjoyment score;
  Min-max values for EEG: 20-100 points.

SECONDARY OUTCOMES:
Awareness of exergame use | Awareness of exergame use was assessed immeditely afterwards exergaming session
  Tool:
  Custom questionnaire aimed to gather detailed information on participants' knowledge and perceptions of exergames as tools for physical training and health improvement.
  Broad range of topics covered aspects such as prior subjects awareness of exergames and VR in physical activity (e.g., "Were you aware that exergames/VR could be used for PA or therapy?"). It also examined participants' opinions on the usefulness of various exergames for physical training (e.g., "Which game do you find most useful for physical training and why?"), and explored their experiences with specific games, such as which left the greatest positive or negative impression. Additionally, questions addressed participants ' current use of modern technologies in PA and their views on how these tools could motivate others in their age group to engage in more PA.
  Scoring: dependently on the question it was adopted Likert scale (in range 1-5), yes/no answer, or multiple answers.
Physical activity | Physical activity was assessed before exergaming session
  Tool:
  International Physical Activity Questionnaire (IPAQ).
  Domains:
  i) vigorous PA - significant effort (rapid breathing and increased heart rate, e.g. running, high-intensity workouts); ii) moderate PA - moderate intensity (slight increase in heart rate, e.g. brisk walking, moderate cycling); iii) walking - all walking during work, transport, or leisure time; iv) sedentary behavior - number of hours spent sitting during a typical day.
  Scoring: Number of MET-minutes/week calculated on the basis of declared time spent on specific activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Poznań University of Physical Education, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 month and ending 3 years after the publication of results
Access Criteria: Who will be able to access the IPD:
  Qualified researchers affiliated with academic or non-profit institutions.
  What will be shared:
  De-identified individual participant data (survey responses and questionnaire scores). Supporting information includes the study protocol and statistical analysis plan.
  How to access the IPD:
  Data will be made available upon reasonable request to the Principal Investigator (PhD Magdalena Cyma-Wejchenig, Poznan University of Physical Education, cyma-wejchenig@awf.poznan.pl). Requests will be reviewed to ensure appropriate use and protection of participant confidentiality.